CLINICAL TRIAL: NCT04878913
Title: Non-interventional, Retrospective, Multicenter, Follow-up Study Evaluating the Effect of C21 on Lung Pathology in Subjects Previously Hospitalized With COVID-19 and Enrolled in the VP-C21-006 Trial
Brief Title: Retrospective Evaluation of Lung Pathology in Subjects With COVID-19
Acronym: ATTRACT-2
Status: Completed | Type: Observational
Sponsor: Vicore Pharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: VP-C21-007
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: COVID-19; COVID-19 Pneumonia
MeSH Terms: conditions — COVID-19 | interventions — compound 21

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C21: Participants treated with C21 in the VP-C21-006 trial
  Interventions: Drug: C21
- Placebo: Participants treated with placebo in the VP-C21-006 trial
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: C21 — C21 was administered in the VP-C21-006 trial
  Other Names: Buloxibutid; Compound 21
  Groups: C21
Drug: Placebo — Placebo was administered in the VP-C21-006 trial
  Groups: Placebo

SUMMARY:
Non-interventional, retrospective, multi-center, follow-up study evaluating the effect of C21 on lung pathology in subjects previously hospitalised with COVID-19 and enrolled in the VP-C21-006 trial.

DETAILED DESCRIPTION:
The study will collect available HRCT scans obtained prior to, during treatment with C21 or placebo and up to 24 weeks after trial completion.

HRCT scans will be assessed for ground glass opacity, reticulation, band opacity, fibrosis and consolidation by a central, blinded HRCT reader.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Previously included in the VP-C21-006 trial and received at least one dose of investigational medicinal product (IMP)
* Available record of at least one HRCT performed within 24 weeks after completion of VP-C21-006.

Exclusion Criteria:

* Participation in another interventional trial during the historical period covered by this study that could interfere with the study objectives or evaluation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who were previously hospitalized with COVID-19 and enrolled in the VP-C21-006 trial.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
Averaged total lung score for both lungs percent measured by per lung percent scores | Up to 24 weeks after completion of VP-C21-006
  Based on ground glass opacity, reticulation, band opacity, fibrosis, and consolidation, on HRCT
Change from baseline in percent lung involvement measured totally (averaged total lung score for both lungs percent) and by each of ground glass opacity, reticulation, band opacity, fibrosis, and consolidation on follow-up HRCT | Up to 24 weeks after completion of VP-C21-006

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Batta, MD, Study Director — Vicore Pharma
Locations (4):
- India (4):
  - Department of Medicine, Civil Hospital and B J Medical College, Ahmedabad, Gujarat
  - First Floor Clinical Research Department Rhythm Heart Institute, Vadodara, Gujarat
  - Department of Medicine, Government Medical College and Hospital, Nagpur, Maharashtra
  - Department of Medicine, Noble Hospitals Pvt. Ltd, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tornling G, et al. The angiotensin type 2 receptor agonist C21 restores respiratory function in COVID19 - a double-blind, randomized, placebo-controlled Phase 2 trial, medRxiv, 2021
- See also: Related Info — https://www.medrxiv.org/content/10.1101/2021.01.26.21250511v1